CLINICAL TRIAL: NCT01573702
Title: Phase II Study of Stereotactic Radiosurgery or Other Local Ablation Followed by Erlotinib for Patients With Epidermal Growth Factor Receptor(EGFR) Mutation Who Have Previously Progressed on an Epidermal Growth Factor Receptor-tyrosine Kinase Inhibitor (EGFR-TKI)
Brief Title: Stereotactic Radiosurgery or Other Local Ablation Then Erlotinib in Epidermal Growth Factor Receptor (EGFR)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 1123
Record Dates: First submitted 2012-04-05; First posted 2012-04-09 (Estimated); Results first posted 2021-01-12 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2020-12

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Non small cell lung cancer; EGFR mutant; Phase II; erlotinib; tarceva; cyberknife; Lineberger
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiosurgery; Erlotinib Hydrochloride

STUDY DESIGN:
Intervention Model Description: For all patients, all sites of progressive disease will be treated with local ablation (primarily stereotactic radiosurgery) followed by the EGFR-TKI erlotinib until disease progression.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stereotactic Radiosurgery Followed by Erlotinib (Other): Stereotactic Radiosurgery or Other Local Ablation Followed by Erlotinib
  Interventions: Procedure: Stereotactic Radiosurgery; Drug: Erlotinib

INTERVENTIONS:
Procedure: Stereotactic Radiosurgery — 21 Gy daily for 5 days
  Other Names: Cyberknife
Drug: Erlotinib — 150mg once daily
  Other Names: Tarceva

SUMMARY:
- Progression free survival after locally ablative therapy and erlotinib in EGFR patients progressed after EGFR-TKI therapy

DETAILED DESCRIPTION:
Primary Objectives

- To estimate progression free survival (PFS) after locally ablative therapy and erlotinib in EGFR-mutant NSCLC patients who progressed on prior EGFR-TKI therapy

Secondary Objectives

* To evaluate local control of sites previously progressive on erlotinib following stereotactic radiosurgery (SRS) followed by erlotinib
* To estimate overall survival (OS) after locally ablative therapy and erlotinib in EGFR-mutant NSCLC patients who progressed on prior EGFR-TKI therapy
* To characterize the toxicity of SRS
* To characterize the toxicity of erlotinib when preceded by SRS

Exploratory Objectives

* To explore if VeriStrat results at initial progression are associated with longer PFS or OS after study treatment
* To explore if VeriStrat results following completion of SRS are associated with longer PFS or OS after re-initiation of erlotinib
* To explore whether "poor" VeriStrat signatures ever turn to "good" signatures with the study therapy, and to explore PFS and OS of patients whose signature changes

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* 18 years of age or older
* Histologically or cytologically confirmed stge IV EGFR-mutant NSCLC
* History of previous response to EGFR-TKI defined by a RECIST 1.1 criteria
* Progressive disease following EGFR-TKI therapy
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Adequate organ and marrow function
* Negative urine or serum pregnancy test for female patients
* Patients who can have children must agree to adequate contraception

Exclusion Criteria:

* Unresolved chronic toxicities greater than 2, measured by CTCAE v4
* Treatment with any FDA approved or experimental cancer treatment following progression on EGFR-TKI
* Any history of previous greater than grade 3 toxicity attributable to erlotinib
* Pregnant or lactating female
* Any previous radiation to sites of planned Stereostatic Radiosurgery
* History of another malignancy
* Concomitant anticancer therapy, immunotherapy, or radiation therapy (within 4 weeks)
* Evidence of severe or uncontrolled systemic diseases
* Known hypersensitivity reaction or idiosyncrasy to erlotinib
* Psychological, familial, sociological, or geographical conditions
* Any other condition in investigator's opinion jeopardize compliance with protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-12-11 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jared Weiss, MD, Principal Investigator — UNC at Chapel Hill
Locations (8):
- United States (8):
  - University of California at San Francisco, San Francisco, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - East Carolina University, Greenville, North Carolina
  - STO Taussig Cancer Center; Cleveland Clinic, Cleveland, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Swedish Cancer Institute, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 32 participants were accrued from six institutions between 12/2012 and 6/2016
Pre-assignment Details: Of the 32 participants who consented to the study, 5 were determined to be not eligible and 2 withdrew consent prior to starting study treatment
Period: Overall Study
Arm/Group | Stereotactic Radiosurgery Followed by Erlotinib
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Stereotactic Radiosurgery Followed by Erlotinib
Number analyzed (Participants) | 25
Age, Continuous [Median (Full Range); unit: years] | 64 [44 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 25
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 25
Smoking status [Count of Participants; unit: Participants]
  Never smoker | 16
  Former smoker | 7
  Unknown | 2
Performance status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status is a scale from 0-5 to describe a patient's level of functioning in terms of self care ability and activity level. Higher on the scale is worse functioning
  Participants
    0, Fully active | 16
    1, Restricted in strenuous activity but ambulatory | 9
Mutation type [Count of Participants; unit: Participants] — The mutation type is the location (Exon) of the mutation in the Epidermal Growth Factor Receptor (EGFR) gene. Subjects who did have proof of a mutation through testing (due to inadequate tissue, for example) were still eligible for the study if they met the clinical criteria of a clinical response overwhelmingly consistent with EGFR mutation (PR plus at least 6 months free of progressive disease as a consequence of EGFR-TKI therapy).
  Participants
    Exon 19 | 14
    Exon 21 | 7
    Exon 19+ ALK rearrangement | 1
    Exon 18 and Exon 20 | 1
    None proven; met clinical criteria | 2
Charlson Co-morbidity Index [Median (Full Range); unit: units on a scale] — The Charlson Comorbidity Index is a method of categorizing comorbidities of patients in which each category has an associated weight (from 1 to 6), based on the adjusted risk of mortality or resource use, and the sum of all the weights results in a single comorbidity score for a patient ranging from 0 (no comorbidities) to 24. The higher the score, the more likely the predicted outcome will result in mortality or higher resource use.
  units on a scale | 6 [0 to 10]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Progression Free Survival
Description: Progression free survival (PFS) after locally ablative therapy and erlotinib in EGFR-mutant NSCLC patients who progressed on prior EGFR-tyrosine kinase inhibitor (TKI) therapy reported as percentage of participants who are alive and without progressive disease at 3 months. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or the appearance of new lesions.
Time Frame: 3 months after Initiation of Stereostatic Radiotherapy
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stereotactic Radiosurgery Followed by Erlotinib
Number analyzed (Participants) | 25
percentage of participants | 64 [42.5 to 82]

2. Secondary Outcome: Percentage of Participants With Local Control of Sites on Erlotinib Following Stereotactic Radiosurgery (SRS)
Description: Count of subjects who had local control of sites previously progressive on erlotinib following SRS followed by erlotinib. Using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), local control is defined as Complete Response (CR), Disappearance of all target lesions; or Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; in sites ablated by SRS.
Time Frame: Initiation of Stereotactic Radiotherapy every 6 to 12 weeks until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
Population: 4 subjects were not evaluable for this outcome due to lack of follow-up measurements on ablated lesions
Measure: Count of Participants; unit: Participants
Arm/Group | Stereotactic Radiosurgery Followed by Erlotinib
Number analyzed (Participants) | 21
Participants | 7

3. Secondary Outcome: Median Overall Survival
Description: To estimate overall survival (OS) after locally ablative therapy and erlotinib in EGFR-mutant, NSCLC patients who progressed on prior EGFR-TKI therapy measured as length of time from start of treatment until date of death from any cause
Time Frame: up to 5 years after end of treatment
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Single Arm Study: Stereotactic Radiosurgery or Other Local Ablation Followed by Erlotinib
  Stereotactic Radiosurgery: 21 Gy daily for 5 days
  Erlotinib: 150mg once daily
Arm/Group | Single Arm Study
Number analyzed (Participants) | 25
Months | 29 [21.7 to 36.3]

4. Secondary Outcome: Toxicity Rate From Stereotactic Radiosurgery (SRS)
Description: Toxicity of SRS will be measured by NCI CTCAE version 4 following completion of SRS, but prior to erlotinib re-initiation. The NCI Common Terminology Criteria for Adverse Events is a descriptive terminology which can be utilized for Adverse Event (AE) reporting. A grading (severity) scale is provided for each AE term. Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental Activities of Daily Living (ADL). Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL. Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE.
Time Frame: From initiation to the end of SRS, up to 15 days
Population: Toxicities occurring in at least two participants from SRS are reported below
Measure: Count of Participants; unit: Participants
Arm/Group | Stereotactic Radiosurgery Followed by Erlotinib
Number analyzed (Participants) | 25
Participants
  Fatigue: Grade 1 | 4
  Fatigue: Grade 2 | 0
  Fatigue: None | 21
  Pain: Grade 1 | 2
  Pain: Grade 2 | 1
  Pain: None | 22
  Anorexia: Grade 1 | 2
  Anorexia: Grade 2 | 0
  Anorexia: None | 23

5. Secondary Outcome: Toxicity Rate Attributed to Erlotinib
Description: Toxicity of erlotinib will be graded using the NCI Common Terminology Criteria for Adverse Events (NCI CTCAE version 4) which is a descriptive terminology which can be utilized for Adverse Event (AE) reporting. A grading (severity) scale is provided for each AE term. Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental Activities of Daily Living (ADL). Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL. Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE.
Time Frame: from end of SRS to end of erlotinib treatment (median duration of 5.7 months)
Population: Toxicities grade 3 or higher and attributed to erlotinib re-treatment, or toxicities occurring in at least two participants are reported below
Measure: Count of Participants; unit: Participants
Arm/Group | Stereotactic Radiosurgery Followed by Erlotinib
Number analyzed (Participants) | 25
Participants
  Acneiform rash: Grade 1 | 5
  Acneiform rash: Grade 2 | 2
  Acneiform rash: Grade 3 | 2
  Acneiform rash: None | 16
  Diarrhea: Grade 1 | 2
  Diarrhea: Grade 2 | 1
  Diarrhea: Grade 3 | 0
  Diarrhea: None | 22
  Fatigue: Grade 1 | 2
  Fatigue: Grade 2 | 1
  Fatigue: Grade 3 | 0
  Fatigue: None | 22
  aspartate aminotransferase (AST) increased: Grade 1 | 2
  aspartate aminotransferase (AST) increased: Grade 2 | 0
  aspartate aminotransferase (AST) increased: Grade 3 | 0
  aspartate aminotransferase (AST) increased: None | 23
  Nausea: Grade 1 | 2
  Nausea: Grade 2 | 0
  Nausea: Grade 3 | 0
  Nausea: None | 23
  Paronychia: Grade 1 | 2
  Paronychia: Grade 2 | 0
  Paronychia: Grade 3 | 0
  Paronychia: None | 23
  Weight loss: Grade 1 | 2
  Weight loss: Grade 2 | 0
  Weight loss: Grade 3 | 0
  Weight loss: None | 23

ADVERSE EVENTS:
Time Frame: From start of treatment to date of death up to 60 months
Arm/Group | Stereotactic Radiosurgery Followed by Erlotinib
All-Cause Mortality (participants affected / at risk) | 16/25
Serious Adverse Events (participants affected / at risk) | 1/25
Other Adverse Events (participants affected / at risk) | 24/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stereotactic Radiosurgery Followed by Erlotinib (N=25)
Fracture (Injury, poisoning and procedural complications) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stereotactic Radiosurgery Followed by Erlotinib (N=25)
Abdominal pain (Gastrointestinal disorders) | 2
Alkaline phosphatase increased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Aspartate aminotransferase increased (Investigations) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 5
Blood bilirubin increased (Investigations) | 1
Blurred vision (Eye disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Bruising (Injury, poisoning and procedural complications) | 1
Conjunctivitis (Eye disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Depression (Psychiatric disorders) | 1
Diarrhea (Gastrointestinal disorders) | 3
Dry eye (Eye disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 4
Dysgeusia (Nervous system disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 3
Dysphagia (Gastrointestinal disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Edema face (General disorders) | 1
Edema limbs (General disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Fatigue (General disorders) | 8
Flashing lights (Eye disorders) | 1
Flu like symptoms (General disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Headache (Nervous system disorders) | 3
Hot flashes (Vascular disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 4
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 1
Infusion site extravasation (General disorders) | 1
Insomnia (Psychiatric disorders) | 1
Lethargy (Nervous system disorders) | 1
Lymphocyte count decreased (Investigations) | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Nail loss (Skin and subcutaneous tissue disorders) | 1
Nail ridging (Skin and subcutaneous tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Neutrophil count decreased (Investigations) | 1
Non-cardiac chest pain (General disorders) | 3
Oral hemorrhage (Gastrointestinal disorders) | 1
Pain (General disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Papulopustular rash (Infections and infestations) | 1
Paronychia (Infections and infestations) | 2
Platelet count decreased (Investigations) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Skin infection (Infections and infestations) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Urinary tract pain (Renal and urinary disorders) | 2
Urinary urgency (Renal and urinary disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Watering eyes (Eye disorders) | 2
Weight loss (Investigations) | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2
White blood cell decreased (Investigations) | 1

LIMITATIONS AND CAVEATS:
The study closed early due to poor accrual (enrolling only 25 of 40 expected participants) and the development of second line therapy with osimertinib.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-11-18): https://cdn.clinicaltrials.gov/large-docs/02/NCT01573702/Prot_SAP_000.pdf